CLINICAL TRIAL: NCT03822780
Title: Hydroxychloroquine in Pediatric ILD With Genetic Surfactant Dysfunction Disorders: Cross-control, Prospective Study
Brief Title: Hydroxychloroquin (HCQ) in chILD of Genetic Defect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jzxfb-qlv
Record Dates: First submitted 2019-01-15; First posted 2019-01-30 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Surfactant Dysfunction
Keywords: Interstitial lung disease; Hydroxychloroquine
MeSH Terms: conditions — Surfactant Dysfunction; Lung Diseases, Interstitial | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: cross-control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCQ Therapy (Experimental): Hydroxychloroquine Sulfate (HCQ, Quensyl) in a loading dose of 10 mg/kg*d, p.o., bid. After the illness gradually alleviate to maintain dose between 5mg/kg*d to 10mg/kg*d, p.o., bid ; the maximum daily dose is 400mg.
  Assess the efficacy and safety of HCQ after 6 months treatment compared with any other routine therapy before HCQ therapy (such as inhaling oxygen, corticosteroid, anti-infection therapy, nutritional support)
  Interventions: Drug: Hydroxychloroquin

INTERVENTIONS:
Drug: Hydroxychloroquin — Hydroxychloroquine Sulfate (HCQ, Quensyl) in a loading dose of 10 mg/kg*d, p.o., bid. After the illness gradually alleviate to maintain dose between 5mg/kg*d to 10mg/kg*d, p.o., bid ; the maximum daily dose is 400mg.
  Other Names: Hydroxychloroquine Sulfate; Plaquenil

SUMMARY:
The purpose of this proposed research is to investigate the efficacy and safety of hydroxychloroquine sulfate (HCQ, Quensyl) for pediatric ILD(chILD) caused by pulmonary surfactant-associated genes mutations.

DETAILED DESCRIPTION:
Children Interstitial lung disease (chILD) is a heterogeneous group of rare respiratory disorders of known and unknown etiologies that are mostly chronic and associated with high morbidity and mortality. ILD are characterized by inflammatory and fibrotic changes of the lung parenchyma structure that typically result in the presence of diffuse infiltrates on lung imaging, and abnormal pulmonary function tests with evidence of a restrictive ventilatory defect and/or impaired gas exchange.

Genetic factors are important contributors to chILD. Genetic variations have been mainly described in genes encoding (or interacting with) the surfactant proteins (SP): SP-C (SFTPC) and the ATP-binding cassette-family A-member 3 (ABCA3) (ABCA3), and less frequently in the genes encoding NKX homeobox 2 (NKX2)-1 (NKX2-1), SP-B (SFTPB), SP-A (SFTPA) and other genes.

To date, the therapeutic managements of such chILD remain limited and are mainly based of the use of corticosteroids, however, their efficacy is highly variable. An alternative approach to treatment was originally described by Tooley who reported a good response to treatment with chloroquine in a girl with ILD, and several case reports have shown a positive response to hydroxychloroquine(HCQ) alone or in combination with systemic steroids of the children with ILD.

The exact mechanism of action of HCQ is unknown, but is probably due to its anti-inflammatory properties, HCQ have lysosomal activities such as diminished vesicle fusion, diminished exocytosis, decreased digestive efficiency of phagolysosomes and reversible "lysosomal storage disease. This may be the mechanism by which HCQ tend to help in chILD, especially in those cases related to surfactant protein deficiency. SP-B and SP-C are synthesized in the endoplasmic reticulum (ER) of alveolar type II cells as large precursor proteins, are cleaved by proteolytic enzymes and transported through Golgi apparatus to multivesicular bodies that fuse with lamellar bodies. In chILD related to SP-C gene mutations, there is misfolding of proSP-C that accumulates within ER and Golgi apparatus in alveolar type II cells, resulting in cellular injury and apoptosis. Treatment with HCQ may interfere with this accumulation of pro-surfactant proteins within alveolar cells.

The investigators propose to study the efficacy and safety of the therapy with HCQ for children with chILD suffered with genetic mutations, and its long-term effects. Through this study the investigators hope to confirm the benefits of HCQ in the treatment of this rare disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be clinically stable for inclusion into the study
* Mature newborn ≥ 37 weeks of gestation, Infants and children (≥2month and < 18y) or previously preterm (≤ 37 weeks of gestation) babies or children(≥2month and <18y) if chILD genetically diagnosed
* chILD genetically diagnosed surfactant dysfunction disorders including patients with mutations in SFTPC, SFTPB, ABCA3, TTF1 (Nkx2-1), FOXF1 further extremely rare entities with specific mutations, for example in TBX4, NPC2, NPC1, NPB, COPA, LRBA and other genes
* no HCQ treatment in the last 3 months
* Ability of subject or/and legal representatives to understand character and individual consequences of clinical trial
* Signed and dated informed consent of the subject (if subject has the ability) and the representatives (of underaged children) must be available before start of any specific trial procedures

Exclusion Criteria:

Subjects presenting with any of the following criteria will not be included in the trial:

* chILD primarily related to developmental disorders
* chILD primarily related to growth abnormalities reflecting deficient alveolarization
* chILD related to chronic aspiration
* chILD related to immunodeficiency
* chILD related to abnormalities in lung vessel structure
* chILD related to organ transplantation/organ rejection/GvHD
* chILD related to recurrent infections
* Acute severe infectious exacerbations
* Known hypersensitivity to HCQ, or other ingredients of the tablets
* Proven retinopathy or maculopathy
* Glucose-6-phosphate-dehydrogenase deficiency resulting in favism or hemolytic anemia
* Myasthenia gravis
* Hematopoetic disorders
* Participation in other clinical trials during the present clinical trial or not beyond the time of 4 half-lives of the medication used, at least one week
* Hereditary galactose intolerance, lactase deficiency or glucose-galactose- malabsorption
* Simultaneous prescription of other potentially nephrotoxic or hepatotoxic medication at the discretion of the treating physician

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Oxygenation change | 6 months
  Clinical judgment of oxygenation condition at 6 months compared with trial day 1 (demand of oxygen supplement while transcutaneous oxygen saturation no less than 92% and with no clinical manifestations of hypoxia)

SECONDARY OUTCOMES:
Oxygen flow rate | 1 month
  O2 supplement(L/min) at 1 months compared with trial day 1
Oxygen flow rate | 3 month
  O2 supplement(L/min) at 3 months compared with trial day 1
Oxygen flow rate | 12 month
  O2 supplement(L/min) at 12 months compared with trial day 1
Oxygen flow rate | 18 month
  O2 supplement(L/min) at 18 months compared with trial day 1
Oxygen flow rate | 24 month
  O2 supplement(L/min) at 24 months compared with trial day 1
Fraction of inspired oxygen(FiO2) | 1 month
  Fraction of inspired oxygen(FiO2) at 1 months compared with trial day 1
Fraction of inspired oxygen | 3 month
  FiO2 at 3 months compared with trial day 1
Fraction of inspired oxygen | 6 month
  FiO2 at 6 months compared with trial day 1
Fraction of inspired oxygen | 12 month
  FiO2 at 12 months compared with trial day 1
Fraction of inspired oxygen | 18 month
  FiO2 at 18 months compared with trial day 1
Fraction of inspired oxygen | 24 month
  FiO2 at 24 months compared with trial day 1
Number of subjects with oxygen inhalation | 6 months
  Number of subjects at 6 months compared with trial day 1
Number of subjects with oxygen inhalation | 12 months
  Number of subjects at 12 months compared with trial day 1
Number of subjects with oxygen inhalation | 24 months
  Number of subjects at 24 months compared with trial day 1
Transcutaneous oxygen saturation | 1 months
  O2-sat at 1 months compared with trial day 1
Transcutaneous oxygen saturation | 3 months
  O2-sat at 3 months compared with trial day 1
Transcutaneous oxygen saturation | 12 months
  O2-sat at 12 months compared with trial day 1
Transcutaneous oxygen saturation | 18 months
  O2-sat at 18 months compared with trial day 1
Transcutaneous oxygen saturation | 24 months
  O2-sat at 24 months compared with trial day 1
Respiratory rate | 1 months
  Respiratory rate(RR) at 1 months compared with trial day 1
Respiratory rate | 3 months
  RR at 3 months compared with trial day 1
Respiratory rate | 6 months
  RR at 6 months compared with trial day 1
Respiratory rate | 12 months
  RR at 12 months compared with trial day 1
Chronic cough | 6 months
  (yes/no)
Chronic cough | 12 months
  (yes/no)
Chronic cough | 24 months
  (yes/no)
Clubbing finger | 6 months
  (yes/no)
Clubbing finger | 12 months
  (yes/no)
Clubbing finger | 24 months
  (yes/no)
Functional lesion of liver and kidney | 3 months
  (yes/no)
Functional lesion of liver and kidney | 6 months
  (yes/no)
Functional lesion of liver and kidney | 12 months
  (yes/no)
Functional lesion of liver and kidney | 24 months
  (yes/no)
Malnutrition | 3 months
  (yes/no) at 3 months compared with trial day 1, based on Reference criteria for growth and development of children under 7 years old in China
Malnutrition | 6 months
  (yes/no) at 6 months compared with trial day 1, based on Reference criteria for growth and development of children under 7 years old in China
Malnutrition | 12 months
  (yes/no) at 12 months compared with trial day 1, based on Reference criteria for growth and development of children under 7 years old in China
Malnutrition | 24 months
  (yes/no) at 24 months compared with trial day 1, based on Reference criteria for growth and development of children under 7 years old in China
Deterioration of pulmonary imaging | 6 months
  (yes/no) Clinical judgment of pulmonary imaging compared with that of last visit if X-ray or CT were done at 6 months
Deterioration of pulmonary imaging | 12 months
  Clinical judgment of pulmonary imaging compared with that of last visit if X-ray or CT were done at 12 months
Deterioration of pulmonary imaging | 24 months
  Clinical judgment of pulmonary imaging compared with that of last visit if X-ray or CT were done at 24 months
Lung function decline | 3 years
  (yes/no) Clinical judgment of Lung-function compared with that of last visit if lung-function testing were done at 3 years
Lung function decline | 6 years
  (yes/no) Clinical judgment of Lung-function compared with that of last visit if lung-function testing were done at 6 years
Abnormal myocardial zymogram | 3 months
  (yes/no)
Abnormal myocardial zymogram | 6 months
  (yes/no)
Abnormal myocardial zymogram | 12 months
  (yes/no)
Duration of oxygen inhalation | 36 months
  The time last from HCQ treatment to withdrawal of oxygen (months)
Mortality | 3 months
  Number of deaths at 3 months
Mortality | 12 months
  Number of deaths at 12 months
Mortality | 24 months
  Number of deaths at 24 months
Number of Treatment related adverse events | 36 months
  Measured on each visit

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Clement A, Nathan N, Epaud R, Fauroux B, Corvol H. Interstitial lung diseases in children. Orphanet J Rare Dis. 2010 Aug 20;5:22. doi: 10.1186/1750-1172-5-22. PMID 20727133
- [Background] Nathan N, Borensztajn K, Clement A. Genetic causes and clinical management of pediatric interstitial lung diseases. Curr Opin Pulm Med. 2018 May;24(3):253-259. doi: 10.1097/MCP.0000000000000471. PMID 29517585
- [Background] Barnett HL. editor. Pediatrics. 15th edition. New York: Appleton Century-Crofts; 1972. pp 1315-1316.
- [Background] Rosen DM, Waltz DA. Hydroxychloroquine and surfactant protein C deficiency. N Engl J Med. 2005 Jan 13;352(2):207-8. doi: 10.1056/NEJM200501133520223. No abstract available. PMID 15647591
- [Background] Kroner C, Reu S, Teusch V, Schams A, Grimmelt AC, Barker M, Brand J, Gappa M, Kitz R, Kramer BW, Lange L, Lau S, Pfannenstiel C, Proesmans M, Seidenberg J, Sismanlar T, Aslan AT, Werner C, Zielen S, Zarbock R, Brasch F, Lohse P, Griese M. Genotype alone does not predict the clinical course of SFTPC deficiency in paediatric patients. Eur Respir J. 2015 Jul;46(1):197-206. doi: 10.1183/09031936.00129414. Epub 2015 Feb 5. PMID 25657025
- [Background] Hevroni A, Goldman A, Springer C. Infant pulmonary function testing in chronic pneumonitis of infancy due to surfactant protein C mutation. Pediatr Pulmonol. 2015 Jun;50(6):E17-23. doi: 10.1002/ppul.23166. Epub 2015 Mar 9. PMID 25755194
- [Background] Avital A, Hevroni A, Godfrey S, Cohen S, Maayan C, Nusair S, Nogee LM, Springer C. Natural history of five children with surfactant protein C mutations and interstitial lung disease. Pediatr Pulmonol. 2014 Nov;49(11):1097-105. doi: 10.1002/ppul.22971. Epub 2013 Dec 17. PMID 24347114
- [Background] Thouvenin G, Abou Taam R, Flamein F, Guillot L, Le Bourgeois M, Reix P, Fayon M, Counil F, Depontbriand U, Feldmann D, Pointe HD, de Blic J, Clement A, Epaud R. Characteristics of disorders associated with genetic mutations of surfactant protein C. Arch Dis Child. 2010 Jun;95(6):449-54. doi: 10.1136/adc.2009.171553. Epub 2010 Apr 19. PMID 20403820
- [Background] Hepping N, Griese M, Lohse P, Garbe W, Lange L. Successful treatment of neonatal respiratory failure caused by a novel surfactant protein C p.Cys121Gly mutation with hydroxychloroquine. J Perinatol. 2013 Jun;33(6):492-4. doi: 10.1038/jp.2012.131. PMID 23719253
- [Background] Arikan-Ayyildiz Z, Caglayan-Sozmen S, Isik S, Deterding R, Dishop MK, Couderc R, Epaud R, Louha M, Uzuner N. Survival of an infant with homozygous surfactant protein C (SFTPC) mutation. Pediatr Pulmonol. 2014 Mar;49(3):E112-5. doi: 10.1002/ppul.22976. Epub 2013 Dec 17. PMID 24347240